CLINICAL TRIAL: NCT05643014
Title: Evaluate the Exposure to Toxicants Emitted During a Structural Fire Assessed by Urinary and Buccal Cell Biomarkers Found in Firefighters.
Brief Title: Observational Study of Exposure to Environmental Toxicants Among Firefighters
Status: Recruiting | Type: Observational
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Responsible Party: Sponsor
Other Study IDs: 2018NTLS135
Record Dates: First submitted 2022-11-30; First posted 2022-12-08 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Healthy
Keywords: PAH; 1-HOP; PheT; SPMA
MeSH Terms: interventions — Specimen Handling

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Participants will provide urine and buccal cell samples.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Firefighters over 18 years old: This is a within subject, observational study of firefighters. This study will involve three sample collections including buccal cells and urine samples; one collection pre and two collections post-structural fire exposure.
  Interventions: Other: Sample collection

INTERVENTIONS:
Other: Sample collection — This study will involve three sample collections including buccal cells and urine samples

SUMMARY:
Observational, within subject study design with 1 pre and 2 post-fire exposure biomarker samples collected to assess exposure to toxicants from combustion emissions related to fighting a structural fire.

ELIGIBILITY:
Inclusion Criteria:

* Firefighter (career or volunteer)
* Over 18 years of age
* Able to provide written voluntary consent

Exclusion Criteria:

* Unwilling to provide a pre and post-exposure urine sample
* Current cancer diagnosis
* Tobacco use within the last 1 year (verified by urinary TNEs)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Firefighters who are exposed to fires containing carcinogens will join this study. Three sample collections will be taken to measure the biomarkers; pre-exposure, 24h post-exposure and 1 week post-exposure.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2020-02-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Studying biomarker levels in firefighters pre and post fire call. | 48 months
  The investigators will evaluate the differences between mean pre-exposure biomarker levels and post-exposure levels in urine and buccal samples collected within 24 hours post-exposure and 1-week post-exposure respectively using t-tests to test for statistical significance.

CONTACTS AND LOCATIONS:
Locations (1):
- Masonic Cancer Center, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Yes
All data will be de-identified and transferred through a secure, password-protected website that is only available to the investigators. All identifying information will be in a locked in a secure place and accessible only to relevant study staff.
Supporting Information: CSR, Analytic Code